CLINICAL TRIAL: NCT02835937
Title: Red Blood Cell Transfusion in the Ambulatory Setting: Impact on Home Functional Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Daryl J. Kor, M.D., Prinicipal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15-006487
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Red Blood Cell Transfusions; Anemia; Hematology; Oncology; Ambulatory Care
MeSH Terms: conditions — Anemia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transfuse (No Intervention): Patients will receive a transfusion under standard care
- No-Transfuse (Experimental): Patients will not receive a transfusion
  Interventions: Other: No-Transfuse

INTERVENTIONS:
Other: No-Transfuse — Patients will not receive an otherwise-indicated red blood cell transfusion
  Arms: No-Transfuse

SUMMARY:
Do ambulatory RBC transfusions improve home functional status?

DETAILED DESCRIPTION:
Background: Red blood cell (RBC) transfusion is frequently employed in both ambulatory and hospital environments with the aim of improving patient functional status. The efficacy of this 10.5 billion dollar per year practice however has been increasingly called into question. The Investigators propose to directly measure the impact of outpatient RBC transfusions on at-home functional status by recording several physiological parameters and quantifiable physical activity metrics, e.g. daily energy expenditure and daily total step count, using the ActiGraph wGT3X-BT. This device is an accelerometer-based wearable similar in size to a small watch and is worn at the waist. Study participants will wear the device during the course of their daily activities giving the investigators quantifiable insight into activity levels in the home environment.

Methods/Design: This will be a randomized crossover pilot clinical trial with participant study duration of 28 days. The crossover nature allows each patient to serve as his/her own control. Details of the study design are provided in the text. Briefly, patients presenting at Mayo Clinic Scottsdale's Ambulatory Infusion Center (AIC) will be randomized to one of two arms: 1) receive an RBC transfusion as scheduled (transfuse), or 2) abstain from the scheduled transfusion (no-transfuse). After an appropriate washout period, patients will cross from the transfuse arm to the no-transfuse arm or vice-versa. Activity levels will be recorded continuously throughout the study with no need for intervention by the patient. In addition to device data, survey data will be collected via a weekly telephone interview. The primary outcome measures will include both technical performance metrics such as daily energy expenditure as well as practical performance metrics such as changes in step count. A variety of secondary outcome measures include daily sedentary time and PROMIS Global 10 scores.

Discussion: This trial will directly assess the impact of red blood cell transfusion on patient functional status in the location most important - the home. Patient recruitment will begin in August 2016 and is due to be completed in August 2017.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* At least on prior encounter in the AIC
* Planned RBC transfusion

Exclusion Criteria:

* Refusal to provide informed consent
* Refusal by the health care team
* Acute ischemia (e.g. MI, CVA)
* Hemoglobin < 7.0 g/dL
* Active bleeding
* Symptomatic anemia (hypotension, tachycardia, angina, syncope/pre-syncope believed related to anemia
* Non-ambulatory functional status
* Established or Uncertain Pregnancy Status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Percent Change in Average Daily Physical Activity | Baseline to 7 Days

CONTACTS AND LOCATIONS:
Overall Officials: Daryl J Kor, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murphree DH, Kinard TN, Khera N, Storlie CB, Ngufor C, Upadhyaya S, Pathak J, Fortune E, Jacob EK, Carter RE, Poterack KA, Kor DJ. Measuring the impact of ambulatory red blood cell transfusion on home functional status: study protocol for a pilot randomized controlled trial. Trials. 2017 Mar 31;18(1):153. doi: 10.1186/s13063-017-1873-z. PMID 28359342